CLINICAL TRIAL: NCT01019382
Title: Phase II Trial of the Effect of Gemcitabine With Intravenous Omega-3 Fish Oil Infusion in Patients With Unresectable Pancreatic Adenocarcinoma
Brief Title: A Study of the Effect of Gemcitabine With Fish Oil in Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Collaborators: B. Braun Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09/H0408/51; EudraCT number 2009-009470027; UHL trial number 10720
Record Dates: First submitted 2009-10-27; First posted 2009-11-25 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Pancreatic Neoplasms
Keywords: pancreatic; carcinoma; cancer; fish; alternative
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma; Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Experimental): All patients entering the trial
  Interventions: Drug: Lipidem fish oil infusion + Gemcitabine chemotherapy

INTERVENTIONS:
Drug: Lipidem fish oil infusion + Gemcitabine chemotherapy — 500mls intravenous infusion once a week of lipidem in addition to standard starting dose of gemcitabine (1000mg/m2) Dose can be reduced if poorly tolerated
  Other Names: Gemzar

SUMMARY:
Over 7000 patients are diagnosed with pancreas cancer every year in the UK. Only 10% have it caught early enough to have surgery to cure it. The rest at best can undergo chemotherapy to extend survival, but current treatments offer at best an improvement of only a few months compared to no treatment at all. In addition only about a quarter of patients will respond to the treatment. In addition these patients often experience profound weight loss, loss of appetite and energy primarily because of the cancer process itself. Our hypothesis is that the addition of fish oil infusion to gemcitabine chemotherapy will result in an improved rate of tumour response on CT imaging.

Fish oils, or specifically the omega-3 fatty acid component, appear to have a range of powerful anti-cancer actions. This is supported by evidence from a wide range of sources, from laboratory experiments to basic human studies. Although this evidence specifically includes many pancreatic cancer studies in the laboratory it has not yet been confirmed in human trials.

Contrary to conventional chemotherapy, fish oil is a naturally occuring non-toxic compound and so is not associated with the side-effects of chemotherapy. In fact a number of clinical studies have demonstrated significant improvements in quality of life for pancreas cancer patients treated with fish oil, particularly with reference to improvements in appetite and energy levels. This is of course in addition to the anti-cancer actions.

DETAILED DESCRIPTION:
Our trial will involve recruiting patients who have unresectable pancreatic cancer and who are suitable for the current standard of care which is gemcitabine chemotherapy. They will be assessed for suitability and then offered entry into the trial. This essentially consists of a 4 hour long infusion of purified omega-3 fish oil immediately after their gemcitabine chemotherapy has finished. This will occur once a week for three weeks, with a rest on the fourth week. The cycle then continues until the cancer has shown progression on a CT scan, the gemcitabine chemotherapy is stopped due to toxicity or the patient withdraws or dies. CT scans to assess this are performed every 2 months. Blood tests will be taken before and after each treatment and analysed for changes in inflammatory markers. The patients will be asked to fill in a quality of life and pain questionnaire each week during the 4 hour infusion.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years
* Able to give informed written consent
* ECOG performance status of 0 or 1 (Appendix 1)
* Life expectancy >12 weeks
* Adequate hepatic and renal function documented within 14 days prior to treatment AST and ALT ≤2.5x upper limit of normal (ULN), unless liver metastases present, in which case ≤5.0xULN Total bilirubin ≤2.5xULN Serum creatinine ≤1.5xULN or calculated creatinine clearance ≥60ml/min Urinary protein <1+ by urine dipstick. If ≥1+, then 24-hour urine collection should be done and may only be enrolled if urine protein is <2g/24hours
* Adequate bone marrow function Haemoglobin ≥9g/dL (can have transfusion or growth factors) Platelets ≥100,000cells/mm3 Neutrophil count ≥1500cells/mm3
* No significant hyperlipidaemia
* Patients without severe blood coagulation disorders (anticoagulants allowed)
* Women of childbearing age must have a negative pregnancy test (urine or serum) at commencement of treatment
* Willingness to comply with scheduled visits, treatment, laboratory test, and other aspects of the trial

Exclusion Criteria:

* Prior treatment with any systemic chemotherapy for metastatic disease
* Prior adjuvant radio- or chemotherapy within 4 weeks of starting the study
* Previous treatment with gemcitabine
* Hypersensitivity to fish-, egg-, or soy protein, or to any of the active substances or constituents in the lipid emulsion
* Any general contra-indications to infusion therapy - pulmonary oedema, hyperhydration, decompensated cardiac insufficiency
* Any unstable medical conditions - uncontrolled diabetes mellitus, acute myocardial infarction, stroke, embolic disease, metabolic acidosis, sepsis, pancreatitis
* Known HIV or AIDS
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with requirements of the protocol
* History of malignancy other than pancreatic cancer, with the exception of curative treatment for skin cancer (other than melanoma) or in situ breast or cervical carcinoma, or those treated with curative intent for any other cancer with no evidence of disease for 5 years
* Major surgical procedure or significant traumatic injury within 4 weeks of treatment
* Female patients must be surgically sterilised or postmenopausal or agree to use two adequate contraception measures during the period of therapy and continued for 6 months after the last dose of gemcitabine. Male patients must be surgically sterilised or agree to use adequate contraception for the same period.
* Patients deemed unsuitable for gemcitabine chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Objective response rate (complete and partial response) on CT according to RECIST criteria | Every 2 months

SECONDARY OUTCOMES:
Overall survival | measured once for each patient
Progression free survival | Measured once for each patient
Safety / tolerability of fish oil and gemcitabine | weekly
Quality of life scores | weekly
brief pain inventory scores | weekly
Pharmacokinetic analysis of blood samples | weekly (before and after treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Dennison, MD FRCS, Principal Investigator — University Hospitals, Leicester; William Steward, Phd FRCP, Study Director — University Hospitals, Leicester; Matthew Metcalfe, MA MD FRCS, Study Chair — University Hospitals, Leicester
Locations (1):
- University Hospitals of Leicester : Leicester Royal Infirmary, Leicester, Leicestershire, United Kingdom

REFERENCES:
- [Background] Park KS, Lim JW, Kim H. Inhibitory mechanism of omega-3 fatty acids in pancreatic inflammation and apoptosis. Ann N Y Acad Sci. 2009 Aug;1171:421-7. doi: 10.1111/j.1749-6632.2009.04887.x. PMID 19723085
- [Background] Chiang KC, Persons KS, Istfan NW, Holick MF, Chen TC. Fish oil enhances the antiproliferative effect of 1alpha,25-dihydroxyvitamin D3 on liver cancer cells. Anticancer Res. 2009 Sep;29(9):3591-6. PMID 19667153
- [Background] Spencer L, Mann C, Metcalfe M, Webb M, Pollard C, Spencer D, Berry D, Steward W, Dennison A. The effect of omega-3 FAs on tumour angiogenesis and their therapeutic potential. Eur J Cancer. 2009 Aug;45(12):2077-86. doi: 10.1016/j.ejca.2009.04.026. Epub 2009 Jun 1. PMID 19493674
- [Background] Funahashi H, Satake M, Hasan S, Sawai H, Newman RA, Reber HA, Hines OJ, Eibl G. Opposing effects of n-6 and n-3 polyunsaturated fatty acids on pancreatic cancer growth. Pancreas. 2008 May;36(4):353-62. doi: 10.1097/MPA.0b013e31815ccc44. PMID 18437081
- [Background] Hering J, Garrean S, Dekoj TR, Razzak A, Saied A, Trevino J, Babcock TA, Espat NJ. Inhibition of proliferation by omega-3 fatty acids in chemoresistant pancreatic cancer cells. Ann Surg Oncol. 2007 Dec;14(12):3620-8. doi: 10.1245/s10434-007-9556-8. Epub 2007 Sep 26. PMID 17896154
- [Background] Merendino N, Loppi B, D'Aquino M, Molinari R, Pessina G, Romano C, Velotti F. Docosahexaenoic acid induces apoptosis in the human PaCa-44 pancreatic cancer cell line by active reduced glutathione extrusion and lipid peroxidation. Nutr Cancer. 2005;52(2):225-33. doi: 10.1207/s15327914nc5202_12. PMID 16201853
- [Background] Shirota T, Haji S, Yamasaki M, Iwasaki T, Hidaka T, Takeyama Y, Shiozaki H, Ohyanagi H. Apoptosis in human pancreatic cancer cells induced by eicosapentaenoic acid. Nutrition. 2005 Oct;21(10):1010-7. doi: 10.1016/j.nut.2004.12.013. PMID 16157238
- [Background] Brown TT, Zelnik DL, Dobs AS. Fish oil supplementation in the treatment of cachexia in pancreatic cancer patients. Int J Gastrointest Cancer. 2003;34(2-3):143-50. doi: 10.1385/IJGC:34:2-3:143. PMID 15361649
- [Derived] Arshad A, Chung WY, Steward W, Metcalfe MS, Dennison AR. Reduction in circulating pro-angiogenic and pro-inflammatory factors is related to improved outcomes in patients with advanced pancreatic cancer treated with gemcitabine and intravenous omega-3 fish oil. HPB (Oxford). 2013 Jun;15(6):428-32. doi: 10.1111/hpb.12002. Epub 2012 Nov 22. PMID 23458624